CLINICAL TRIAL: NCT01171534
Title: Closure of Fasciotomy Wounds: A Prospective, Observational Study of a Continuous External Tissue Expander
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study determined not to be feasible to continue.
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Wound Care Technologies, Inc. (Industry)
Responsible Party: Principal Investigator, Gregory Della Rocca, Associate Professor, Co-Director of Trauma Services, Department of Orthopaedic Surgery, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB1162817
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Results first posted 2014-12-10 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Wounds and Injuries; Compartment Syndrome
MeSH Terms: conditions — Wounds and Injuries; Compartment Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vessel Loop fasciotomy closure (Active Comparator): Fasciotomy closure using vessel loops and staples.
  Interventions: Device: Vessel loop
- DermaClose fasciotomy closure (Experimental): Fasciotomy closure via DermaClose device
  Interventions: Device: DermaClose fasciotomy closure

INTERVENTIONS:
Device: DermaClose fasciotomy closure — The DermaClose device provides continuous expanding of the skin around the wound until it has stretched enough to allow the skin edges to be sutured closed.
  Other Names: Continuous External Tissue Expander
  Arms: DermaClose fasciotomy closure
Device: Vessel loop — Vessel loops and staples for fasciotomy closure
  Arms: Vessel Loop fasciotomy closure

SUMMARY:
Fasciotomy wounds are rarely able to be closed at the time of index surgery. They often require multiple returns to surgery for closure, and occasionally require skin grafting (i.e. they are never completely closed). We are interested in seeing whether this device, which provides constant and gradual tension on the wound, may allow for rapid wound closure in a safe fashion, perhaps even precluding a return trip to surgery.

Null hypothesis #1: The Dermaclose Wound Management System (Woundcare Technologies Inc, Chanhassen, Minnesota) will not result in closure of fasciotomy wounds more rapidly than standard vessel loop techniques.

Null hypothesis #2: The Dermaclose Wound Management System will not reduce the number of return trips to the operating room for surgical procedures related to closure or skin grafting of fasciotomy wounds.

DETAILED DESCRIPTION:
After IRB approval, all patients meeting inclusion criteria and requiring fasciotomy of the arms, legs, or pelvis will be consented for participation in the research study. Patients will either have their fasciotomy wounds closed through application of the Dermaclose device, as per the manufacturer's instructions, or through application of vessel loops with staples in a "shoestring technique" as described in the literature (1). Choice of wound closure technique will be at surgeon discretion. All patients will undergo application of a vacuum-assisted wound closure device (Wound VAC, Active Healing Solutions Inc, San Antonio, TX), which is standard of care for temporary coverage of open wounds (2, 3). Patients will be returned to the operating room every 2-3 days until wound closure or skin grafting has been accomplished. If skin closure is not accomplished in the operating room, but occurs prior to return trip to the operating room, then definitive suture closure of the wound will be performed under local anaesthetic, followed by removal of the Dermaclose device or of the vessel loop with staple shoestring. Decisions regarding wound closure or skin grafting in the operating room will be left to the judgment of the attending surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients undergoing fasciotomy for decompression of compartment syndrome, evolving compartment syndrome, or prophylactically to prevent compartment syndrome

Exclusion Criteria:

* Patient younger than 18 years of age
* Patients with an active infection
* Patients unable to comply with protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-07; Primary Completion 2013-08 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Della Rocca, MD. PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Hospital and Clinics, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- DermaClose Fasciotomy Closure: Fasciotomy closure via DermaClose device
  DermaClose Continuous External Tissue Expander: The DermaClose device provides continuous expanding of the skin around the wound until it has stretched enough to allow the skin edges to be sutured closed.
Period: Overall Study
Arm/Group | Vessel Loop Fasciotomy Closure | DermaClose Fasciotomy Closure
Started | 0 (retrospective arm never performed on study) | 7
Completed | 0 | 4
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — screen failure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vessel Loop Fasciotomy Closure | DermaClose Fasciotomy Closure | Total
Number analyzed (Participants) | 0 | 7 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 7 | 7
  >=65 years |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 7 | 7

OUTCOME MEASURES:

1. Primary Outcome: Performance of DermaClose System in Treatment of Fasciotomy Wounds
Description: Days to wound closure; number and types of procedures required for wound closure; infection requiring reoperation; wound dehiscence requiring reoperation
Time Frame: One year
Population: Too low of an enrollment volume to analyze
Arm/Group | Vessel Loop Fasciotomy Closure | DermaClose Fasciotomy Closure
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Pain
Description: Visual Analog Pain Scale (VAS) during initial hospitalization and at 2 weeks, 6 weeks, 3 months, 6 months, and 12 months
Time Frame: One Year
Population: too low of an enrollment volume to analyze
Arm/Group | Vessel Loop Fasciotomy Closure | DermaClose Fasciotomy Closure
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Quality of Life
Description: Quality of Life measured by the SF-12 version 1 at 2 weeks, 6 weeks, 3 months, 6 months, and 12 months
Time Frame: One Year
Population: This study was terminated before any of this information was collected and analyzed.
Arm/Group | Vessel Loop Fasciotomy Closure | DermaClose Fasciotomy Closure
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Cost-to-Benefit Ratio of DermaClose Versus Vessel Loop Fasciotomy Closure
Description: Costs associated with both types of closure (DermaClose and Vessel Loop) including hospital days, number of procedures, procedural and hospital costs including device(s), negative pressure wound therapy costs, and operating room time and associated costs.
Time Frame: One year
Population: This study was terminated before this information was collected and analyzed.
Arm/Group | Vessel Loop Fasciotomy Closure | DermaClose Fasciotomy Closure
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Vessel Loop Fasciotomy Closure | DermaClose Fasciotomy Closure
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/7
Other Adverse Events (participants affected / at risk) | 0/0 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less